CLINICAL TRIAL: NCT07337174
Title: A Randomized, Open-label, Single Dose, Two-way, Crossover, Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetics After Subcutaneous Injection of HUC2-676 or HUC2-676-R in Healthy Adult Subjects
Brief Title: Study to Compare and Evaluate the Safety and Pharmacokinetics After Subcutaneous Injection of HUC2-676 or HUC2-676-R in Healthy Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUC2-676
Record Dates: First submitted 2025-12-22; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUC2-676 (Experimental)
  Interventions: Drug: HUC2-676
- HUC2-676-R (Active Comparator)
  Interventions: Drug: HUC2-676-R

INTERVENTIONS:
Drug: HUC2-676 — subcutaneous injection
  Arms: HUC2-676
Drug: HUC2-676-R — subcutaneous injection
  Arms: HUC2-676-R

SUMMARY:
The trial uses a randomized, open-label, single-dose administration per period, and a 2 x 2 crossover design where subjects receive both treatments sequentially with a washout.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19 to 65 years, inclusive, at screening.
* Subjects who have been fully informed of the details of this clinical trial, have fully understood the information, have voluntarily decided to participate, and have provided written informed consent to comply with all protocol requirements throughout the trial period.

Exclusion Criteria:

* Subjects with a current or past clinically significant medical history of hepatic, renal, neurological, psychiatric, respiratory, endocrine, hematologic, oncologic, genitourinary, cardiovascular, gastrointestinal, musculoskeletal, or other disorders.
* For females: Pregnant women (positive urine hCG) or nursing mothers.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Cmax following single-dose administration | 0 through 72 hours post-dose
AUC following single-dose administration | 0 through 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Park, Principal Investigator — Chungbuk National University Hospital

IPD SHARING:
Plan to Share IPD: No